CLINICAL TRIAL: NCT01807819
Title: The Determination of Important Mechanical Patterns of Left Ventricular Efficiency-MV02 Study
Acronym: DIMPLE
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201602538; 27-2013 (Other: uf legacy)
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure
Keywords: Heart Failure; Myocardial Strain; Functional Capacity
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure: Patients will undergo echocardiogram and exercise testing. Two year phone follow-up.
  Interventions: Other: Heart Failure

INTERVENTIONS:
Other: Heart Failure — Patients will undergo echocardiogram and exercise testing. Two year phone follow-up.

SUMMARY:
The purpose of this study is to determine if analysis of heart ultrasound images with new software programs will provide better understanding as to the specific heart problems that lead to symptoms of heart failure.

DETAILED DESCRIPTION:
1. Research Plan:

   Patients: Patients 18 years of age or older who are referred to our adult cardiovascular Echocardiograms: Patients will have a focused echocardiogram performed in the Cardiovascular Clinic at rest and immediately after symptom limited treadmill stress. Echocardiograms will be obtained in the left lateral decubitus position with an iE33 (Philips, The Netherlands) machine equipped with a broadband S5-1 transducer (frequency transmitted 1.7MHz, received 3.4 MHz). Parasternal long- and short axis views will be obtained at the basal (tips of the mitral valve visualized), midventricular (papillary muscles visualized) and apical levels (just proximal to the level of end-systolic LV luminal obliteration, with the transducer positioned 1 or 2 intercostal spaces more caudal to allow the LV to be viewed as circular as possible). Additionally, three standard apical views (4-chamber, 2-chamber, and 3-chamber) will be obtained. To optimize speckle tracking, images will be acquired at as high as a frame rate as possible (50-90 frames/s) and every effort will be made for the endocardial and epicardial border to be visualized throughout the cardiac cycle. Pulsed wave Doppler will be acquired at the level of the mitral valve leaflet tips, and at the pulmonary vein as seen from the apical 4-chamber view. A color Doppler M-mode image including the LV apex and the open mitral valve will be obtained with the upper Nyquist limit set to 45cm/sec. Tissue Doppler velocities will be acquired at the medial and lateral mitral annulus.

   Echocardiogram Analysis: All data analysis will be performed by an investigator masked to the patient's history and peak VO2 and 6 minute walk results. LV end-systolic and end-diastolic volumes and ejection fraction will be determined by manual tracing of the end-systolic and end-diastolic endocardial borders using apical 4- and 2-chamber views, employing Simpson's biplane method. Pulsed wave Doppler at the level of the mitral valve leaflet tips will be used to determine peak early (E) and atrial (A) filling velocities, and deceleration time (DT). Tissue Doppler will be used to determine peak early (E') velocity of the medial and lateral mitral annulus. The LV apical color M Mode image will be used to determine the propagation velocity.

   Speckle Tracking Analysis: Analyses will be performed using QLAB advanced quantification software version 7.1 (Philips, The Netherlands). Short axis and long axis images will be automatically divided into six segments. Automated tracking of myocardial speckles will be reviewed and manually adjusted as minimally as possible. The tracking quality of each segment will be visually evaluated and if tracking is felt to be inaccurate, strain analysis of that segment will not be included. Speckle tracking analysis provides peak and time to peak measures of circumferential, radial and longitudinal strain in 18 LV segments. Additionally, speckle tracing analysis provides peak and time to peak measures of bulk, endocardial and epicardial twist in the basal, mid, and apical LV regions. If less than 2/3 of the components for a computed variable are available, than that computed variable will not be included in the relevant analysis.

   Graded exercise testing for assessment of peak oxygen consumption (Stress Protocol): We will use a Naughton-Balke treadmill protocol where the speed will be kept at 3.0 mph and the grade will be increased 2.5% every 2 minutes- a modified protocol using 2.0 mph will be adopted for slow walkers. A valid test will be defined according to the ATS/ACCP statement on cardiopulmonary exercise testing as meeting at least one of the following criteria: Plateau in VO2, heart rate (HR) within 10 beats/min of age-predicted maximal HR, respiratory exchange ratio > 1.10, exhaustion defined as RPE of 9-10 on the Borg CR-10 scale, or achievement of predicted maximal work rate. Patients will be verbally encouraged before and during the test, to give a maximal effort with the goal of achieving physiological limitation. Criteria for exercise termination will include: chest pain suggestive of ischemia, ischemic ECG changes, complex ectopy, second or third degree heart block, fall in systolic blood pressure >20mmHg from highest value during the test, hypertension (>250 mmHg systolic; >120 diastolic), severe desaturation: SpO2 < 80% when accompanied by symptoms and signs of severe hypoxemia, sudden pallor, loss of coordination, mental confusion, dizziness or faintness, signs of respiratory failure. In situations in which the test is prematurely terminated the patient will be observed until they are stable and physiologic variables have returned to baseline conditions. If necessary and based on the criteria of the physician, admission to the hospital may be warranted. Resuscitation (i.e. crash cart) equipment will be available in the laboratory for such occurrences.

   Quantification of peak oxygen consumption: Oxygen consumption will be measured using a portable Cosmed K4b2. The Cosmed K4b2 weighs 1.5 kg, including the battery and specially designed harness and has been validated against Douglas bags during steady-state exercise. The mass of this device will be added to total body mass in calculating peak oxygen consumption in ml/kg/min. Oxygen consumption will be measured breath-by-breath and subsequently averaged over 10-second periods. Participants will be asked not to talk during testing and will be instructed to use hand signals to communicate with the research assistants. Heart rate will be measured simultaneously during all tasks using a Polar heart rate monitor (Model RS100, Polar Electro Inc.). As of October 2015 functional capacity will be evaluated with 6 minute walk test.
2. Possible Discomforts and Risks:

   The major risk being undertaken in this study is cardiopulmonary exercise testing. In general, maximal symptom-limited exercise testing is a relatively safe procedure. In a survey of 1,375 clinical exercise testing facilities, the risk of dying during the cardiopulmonary exercise test was 0.5 per 10,000 tests. It is important to understand that exercise is performed outside of a clinic setting on a regular basis without supervision. We will take every measure possible to limit the risk of exercise to study participants. We will conduct a thorough medical examination and review the resting ECG prior to exercise. Those patients with contraindication to exercise testing will not exercise and will not continue in this study. Additionally, we will continuously monitor 12-lead ECGs during exercise to check for signs of myocardial ischemia. A fully equipped crash cart is available if an event were to occur. All treadmill testing will be conducted under the supervision of a physician and/or appropriately trained nurse practitioners. The nurse practitioner will be trained and certified in exercise testing. All testing supervisors have a thorough knowledge of normal and abnormal exercise responses and are certified in cardiac life support. They will be able to recognize an abnormal rhythm and ST depression on an electrocardiogram. All sites have on-call access to a study physician and contact numbers for emergency services. Institutional and community EMS services will be activated if needed.
3. Possible Benefits:

There are no possible benefits to the health of the patient during study. Discoveries made during the investigation could potentially benefit the study participants or other patients with cardiovascular disease in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older who are referred to our adult cardiovascular heart failure clinics for evaluation of heart failure or LV dysfunction.

Exclusion Criteria:

* Patients with contraindications to exercise testing:(myocardial infarction within 2 days, unstable angina, uncontrolled cardiac arrhythmias, severe aortic stenosis, uncontrolled symptomatic heart failure, recent pulmonary embolism, recent myocarditis, history of aortic dissection, untreated ischemic CAD, blood pressure > 200/110, history of untreated tachy- or brady arrhythmia, hypertrophic cardiomyopathy, or inability to perform exercise because of physical or mental impairment) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who are referred to our adult cardiovascular heart failure clinics for evaluation of heart failure or LV dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Correlation of myocardial strain with maximal oxygen consumption | Baseline

SECONDARY OUTCOMES:
Cardiovascular Hospitalization | Baseline to 2 years
Cardiovascular Death | Baseline to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John W Petersen, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Shands Cardiovascular Clinic, Gainesville, Florida, United States